CLINICAL TRIAL: NCT05347095
Title: A Phase 3, Randomized, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of Guselkumab in Participants With Fistulizing, Perianal Crohn's Disease
Brief Title: A Study of Guselkumab in Participants With Fistulizing, Perianal Crohn's Disease
Acronym: FUZION CD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109189; CNTO1959CRD3005 (Other: Janssen Research & Development, LLC); 2021-000491-10 (EudraCT Number); 2023-504740-33-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Fistulizing Crohns Disease; Perianal Crohns Disease
MeSH Terms: interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Guselkumab (Experimental): Participants will receive guselkumab Dose 1 intravenous (IV) infusion followed by Dose 2 subcutaneously (SC). Participants will receive matching placebo to maintain the blind. Participants who are eligible and willing to continue guselkumab may enter the Long-Term Extension (LTE) period and continue to receive guselkumab.
  Interventions: Drug: Guselkumab; Drug: Placebo
- Group 2: Guselkumab (Experimental): Participants will receive guselkumab Dose 1 IV infusion followed by Dose 3 SC. Participants will receive matching placebo to maintain the blind. At Week 24, guselkumab Dose 3 SC non-responders will switch to receive guselkumab dose 2 SC. Participants who are eligible and willing to continue guselkumab may enter the LTE period and continue to receive guselkumab.
  Interventions: Drug: Guselkumab; Drug: Placebo
- Group 3: Placebo (Experimental): Participants will receive placebo IV infusion followed by placebo SC. At Week 24, placebo non-responders will continue to receive guselkumab Dose 4 followed by guselkumab Dose 2 SC. Participants will receive matching placebo to maintain the blind. Participants who are eligible and willing to continue guselkumab may enter the LTE period and continue to receive guselkumab.
  Interventions: Drug: Guselkumab; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered subcutaneously/IV infusion.
  Other Names: CNTO1959
Drug: Placebo — Matching placebo will be administered subcutaneously/IV infusion.

SUMMARY:
The purpose of this study to evaluate the clinical efficacy of guselkumab in fistulizing, perianal Crohn's disease and to assess the overall safety of guselkumab.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of Crohn's disease with a minimum duration of at least 3 months
* Has at least one active draining perianal fistula as a complication of Crohn's disease, confirmed by screening magnetic resonance imaging (MRI) results
* Has previously demonstrated lack of initial response (that is primary non-responders), responded initially but then lost response with continued therapy (that is secondary non-responders), or were intolerant to a maximum of 2 classes of advanced drug therapies at a dose approved for the treatment of Crohn's disease (that is infliximab, adalimumab, certolizumab pegol, vedolizumab, or approved biosimilars for these agents) or JAK inhibitors licensed for Crohn's disease treatment (that is, upadacitinib)

Exclusion Criteria:

* Has a very severe luminal disease activity
* History of concurrent rectovaginal fistulas (other types of concurrent fistula should be confirmed with the sponsor), rectal and/or anal stenosis, stoma or functioning ostomy (include all current stoma types abscess or collections which are not properly drained) colonic mucosal dysplasia or pre-cancerous lesions that have not been removed, demyelinating disease, or systemic lupus erythematosus
* Has complications of CD, such as symptomatic strictures or stenoses, short gut syndrome, or any other manifestation that might be anticipated to require surgery or preclude fistula evaluation
* Any medical contraindications preventing study participation
* Has a history of ongoing, chronic or recurrent enteral or systemic infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2027-03-25 (Estimated); Study Completion 2027-03-25 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Combined Fistula Remission at Week 24 | Week 24
  Percentage of participants who achieve combined fistula remission at Week 24 will be reported. Combined fistula remission is defined as 100 percentage (%) closure of all treated external openings without development of new fistulas or abscesses and without any drainage by the external openings [occurring spontaneously or after gentle finger compression] and absence of collections greater than (>) 2 centimeters (cm) of the perianal fistulas in at least two of three dimensions, confirmed by a blinded central review of the magnetic resonance imaging [MRI] results.

SECONDARY OUTCOMES:
Percentage of Participants who Achieve Combined Fistula Remission at Week 48 | Week 48
  Percentage of participants who achieve combined fistula remission at Week 48 will be reported.
Percentage of Participants who Achieve Clinically Assessed Fistula Remission | Week 24
  Percentage of participants who achieve clinically assessed fistula remission will be reported. Clinically assessed fistula remission is defined as 100% closure of all treated external openings, without development of new fistulas or abscesses and without any drainage by the external openings, occurring spontaneously or after gentle finger compression.
Percentage of Participants who Achieve Radiological Fistula Remission Based on Radiological Findings Assessed by MRI | Week 24
  Percentage of participants who achieve radiological fistula remission based on radiological findings assessed by MRI will be reported. Radiological remission is defined as absence of collections >2 cm of the perianal fistulas in at least two of three dimensions, confirmed by a blinded central review of the MRI results.
Percentage of Participants who Achieve Clinically Assessed Fistula Response at Week 24 | Week 24
  Percentage of participants who achieve clinically assessed fistula response at Week 24 will be reported. Clinically assessed fistula response is defined as a greater than or equal to (>=) 50% reduction from baseline in number of open or draining perianal fistulas.
Percentage of Participants who Achieve Clinically Assessed Fistula Response at Week 12 | Week 12
  Percentage of participants who achieve clinically assessed fistula response at Week 12 will be reported. Clinically assessed fistula response is defined as >=50% reduction from baseline in number of open or draining perianal fistulas.
Change from Baseline in Crohn's Disease Activity Index (CDAI) by Visit Over Time Through Week 48 | Baseline up to Week 48
  Change from baseline in CDAI by visit over time will be reported. CDAI will be assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid or very soft stools, abdominal pain (AP)/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being with scores ranging from 0 to approximately 600. The last 4 variables are scored over 7 days by the participant on a diary card that participants are to complete on a daily basis.
Percentage of Participants who Achieve Clinical Remission (CDAI less than [<] 150) by Visit Over Time Through Week 48 Among Participants with CDAI Greater than (>) 150 at Baseline | Through Week 48
  Percentage of participants who achieve clinical remission (CDAI <150) by visit over time through Week 48 among participants with CDAI >150 at baseline will be reported. CDAI will be assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid or very soft stools, abdominal pain [AP]/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being with scores ranging from 0 to approximately 600. The last 4 variables are scored over 7 days by the participant on a diary card that participants are to complete on a daily basis.
Percentage of Participants who Achieve a Clinical Response by Visit Over Time Through Week 48 Among Participants with CDAI >150 at Baseline | Through Week 48
  Percentage of participants who achieve a clinical response by visit over time through Week 48 among participants with CDAI >150 at baseline will be reported. Clinical response is defined greater than or equal to (>=) 100-point reduction from baseline in CDAI, or CDAI <150.
Percentage of Participants who Achieve Steroid-free Clinical Remission by Visit Over Time Through Week 48 Among Participants with CDAI >150 at Baseline | Through Week 48
  Percentage of participants who achieve steroid-free clinical remission by visit over time through Week 48 among participants with CDAI >150 at baseline will be reported. Steroid-free clinical remission is defined as CDAI <150 and not receiving corticosteroids by visit over time through Week 48 among participants with CDAI >150 at baseline.
Percentage of Participants who Achieve Combined Clinical Response and Clinically Assessed Fistula Response Among Participants With CDAI >220 at Baseline | Week 24 and Week 48
  Percentage of participants who achieve combined clinical response and clinically assessed fistula response among participants with CDAI >220 at baseline at baseline will be reported. Clinical response is defined >=100-point reduction from baseline in CDAI, or CDAI <150. Clinically assessed fistula response is defined as >=50% reduction from baseline in number of open or draining perianal fistulas.
Percentage of Participants who Achieve Combined Clinical Remission and Clinically Assessed Fistula Remission Among Participants with CDAI >220 at Baseline | Week 24 and Week 48
  Percentage of participants who achieve combined clinical remission and clinically assessed fistula remission among participants with CDAI >220 at baseline at will be reported. Clinical remission is defined as CDAI <150. Clinically assessed fistula remission is defined as 100% closure of all treated external openings, without development of new fistulas or abscesses and without any drainage by the external openings, occurring spontaneously or after gentle finger compression.
Percentage of Participants who Achieve Combined Clinical Response and Clinically Assessed Fistula Remission Among Participants with CDAI >220 at Baseline | Week 24 and Week 48
  Percentage of participants who achieve combined clinical response and clinically assessed fistula remission among participants with CDAI >220 at baseline will be reported. Clinical response is defined >=100-point reduction from baseline in CDAI, or CDAI <150. Clinically assessed fistula remission is defined as 100% closure of all treated external openings, without development of new fistulas or abscesses and without any drainage by the external openings, occurring spontaneously or after gentle finger compression.
Percentage of Participants who Achieve Combined Clinical Remission and Clinically Assessed Fistula Response among Participants with CDAI >220 at Baseline | Week 24 and Week 48
  Percentage of participants who achieve combined clinical remission and clinically assessed fistula response among participants with CDAI >220 at baseline will be reported. Clinically assessed fistula response is defined as >=50% reduction from baseline in number of open or draining perianal fistulas.
Percentage of Participants who Achieve Combined Clinical Response and Clinically Assessed Fistula Response at Week 24 and Week 48 | Week 24 and Week 48
  Percentage of participants who achieve combined clinical response and clinically assessed fistula response at Week 24 and Week 48 will be reported. Clinical response is defined >=100-point reduction from baseline in CDAI, or CDAI <150. Clinically assessed fistula response is defined as >=50% reduction from baseline in number of open or draining perianal fistulas.
Percentage of Participants who Achieve Combined Clinical Response and Clinically Assessed Fistula Remission at Week 24 and Week 48 | Week 24 and Week 48
  Percentage of participants who achieve combined clinical response and clinically assessed fistula remission at Week 24 and Week 48 will be reported. Clinical response is defined >=100-point reduction from baseline in CDAI, or CDAI <150. Clinically assessed fistula remission is defined as 100% closure of all treated external openings, without development of new fistulas or abscesses and without any drainage by the external openings, occurring spontaneously or after gentle finger compression.
Percentage of Participants who Achieve Combined Clinical Remission and Clinically Assessed Fistula Response at Week 24 and Week 48 | Week 24 and Week 48
  Percentage of participants who achieve combined clinical remission and clinically assessed fistula response at Week 24 and Week 48 will be reported. Clinically assessed fistula response is defined as >=50% reduction from baseline in number of open or draining perianal fistulas.
Percentage of Participants who Achieve Combined Clinical Remission and Clinically Assessed Fistula Remission at Week 24 and Week 48 | Week 24 and Week 48
  Percentage of participants who achieve combined clinical remission and clinically assessed fistula remission will be reported. Clinically assessed fistula remission is defined as 100% closure of all treated external openings, without development of new fistulas or abscesses and without any drainage by the external openings, occurring spontaneously or after gentle finger compression.
Change from Baseline in Perianal Disease Activity Index (PDAI) Overall Score, Discharge Score, and Pain Score by Visit Over Time Through Week 48 | Baseline up to Week 48
  Change from baseline in PDAI overall score, discharge score, and pain score by visit over time through Week 48 will be reported. The PDAI is a scoring system to evaluate the severity of perianal lesion associated with Crohn's disease. It includes the following 5 items: (a) Discharge; (0=no discharge to 4= Gross fecal soiling) (b) Pain; (0=no activity to 4= severe pain, severe limitation) (c) Restriction of sexual activity;(0=no perianal disease/skin tags to 4= unable to engage in sexual activity) (d) Type of perianal disease; (0=no perianal disease/skin tags to 4=Anal sphincter ulceration or fistulae with significant undermining ok skin) and (e) Degree of induration; (0=no induration to 4=gross fluctuance/abscess. Higher scores indicate more severe or active disease.
Percentage of Participants who Achieve Clinically Assessed Fistula Response by Visit Over Time Through Week 48 | Through Week 48
  Percentage of participants with clinically assessed fistula response by visit over time through Week 48 will be reported. Clinically assessed fistula response is defined as >=50% reduction from baseline in number of open or draining perianal fistulas.
Percentage of Participants who Achieve Clinically Assessed Fistula Remission by Visit over Time Through Week 48 | Through Week 48
  Percentage of participants with clinically assessed fistula remission by visit over through Week 48 time will be reported. Clinically assessed fistula remission is defined as 100% closure of all treated external openings, without development of new fistulas or abscesses and without any drainage by the external openings, occurring spontaneously or after gentle finger compression.
Percentage of Participants who Achieve Clinically Assessed Fistula Remission at Week 48 Among the Participants who Achieve Clinical Fistula Remission at Week 24 | Week 48
  Percentage of participants who achieve clinically assessed fistula remission at Week 48 among the participants who achieve clinical fistula remission at Week 24 will be reported. Clinically assessed fistula remission is defined as 100% closure of all treated external openings, without development of new fistulas or abscesses and without any drainage by the external openings, occurring spontaneously or after gentle finger compression.
Percentage of Participants who Achieve Clinically Assessed Fistula Remission at Week 48 Among Those who Achieve Fistula Remission or Response at Week 24 | Week 48
  Percentage of participants achieving clinically assessed fistula remission at Week 48 among those who achieve fistula remission or response (defined either by clinical or radiological assessment) at Week 24 will be reported. Clinically assessed fistula remission is defined as 100% closure of all treated external openings, without development of new fistulas or abscesses and without any drainage by the external openings, occurring spontaneously or after gentle finger compression.
Time to Clinical Fistula Remission | Up to Week 96
  Time to clinical fistula remission will be reported. Clinical fistula remission is defined as 100% closure of all treated external openings without development of new fistulas or abscesses and without any drainage by the external openings (occurring spontaneously or after gentle finger compression).
Percentage of Participants who Achieve Radiological Fistula Predominantly Fibrotic Status for all Existent Fistulas Assessed by MRI at Week 24 and Week 48 | Week 24 and Week 48
  Percentage of participants who achieve radiological fistula predominantly fibrotic status for all existent fistulas assessed by MRI at Week 24 and Week 48 will be reported.
Percentage of participants who Achieve Radiological Remission Based on Radiological Findings Assessed by MRI at Week 48 | Week 48
  Percentage of participants with radiological remission based on radiological findings assessed by MRI at Week 48 will be reported. Radiological remission is defined as absence of collections >2 cm of the perianal fistulas, confirmed by a blinded central review of the MRI results.
Percentage of Participants who Achieve Radiological Remission Assessed by MRI at Week 48 Among the Participants who Achieve Radiological Remission at Week 24 | Week 48
  Percentage of participants who achieve radiological remission assessed by MRI at Week 48 among the participants who achieve radiological remission at Week 24 will be reported. Radiological remission is defined as absence of collections >2 cm of the perianal fistulas, confirmed by a blinded central review of the MRI results.
Percentage of Participants who Achieve Combined Clinically Assessed and Radiological Fistula Remission at Week 48 Among the Participants who Achieve Combined Clinical and Radiological Fistula Remission at Week 24 | Week 48
  Percentage of participants who achieve combined clinically assessed and radiological (assessed by MRI) fistula remission at Week 48 among the participants who achieve combined clinical and radiological fistula remission at Week 24.
Percentage of Participants who Achieve Combined Clinically Assessed and Radiological Fistula Remission at Week 48 Among the Participants with Clinical Fistula Response at Week 24 | Week 48
  Percentage of participants who achieve combined clinically assessed and radiological (assessed by MRI) fistula remission at Week 48 among the participants who achieve clinical fistula response at Week 24 will be reported.
Percentage of Participants with Proctitis at Week 48 Among Participants with MRI-confirmed Proctitis at Baseline | Week 48
  Percentage of participants with proctitis at Week 48 among participants with MRI-confirmed proctitis at baseline will be reported. Proctitis is defined as the inflammation of the lining of the rectum.
Change from Baseline in Magnetic Resonance Novel Index for Fistula imaging in Crohn's disease (MAGNIFI-CD) by Visit Over Time Through Week 48 | Baseline up to Week 48
  Change from baseline in MAGNIFI-CD by visit over time through Week 48 will be reported. The MAGNIFI-CD is based on MRI assessment of 6 items including number of fistula tracts, fistula length, hyperintensity of primary tract on post-contrast T1-weighted images, dominant feature, extension, and inflammatory mass. The total MAGNIFI-CD score ranges from 0 (no disease activity) to 25 (severe disease activity). It assesses the MRI data and determines perianal fistulizing CD activity with improved operating characteristics compared to the Van Assche Index (VAI) and the modified VAI (mVAI).
Change from Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) by Visit Over Time Through Week 48 | Baseline up to Week 48
  Change from baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) by visit over time through Week 48 will be reported. The IBDQ is a validated, 32-item, self-reported questionnaire for participants with IBD to evaluate patient reported outcomes (PROs) across 4 dimensions: bowel symptoms (loose stools, AP), systemic symptoms (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability). Scores range from 32 to 224, with higher scores indicating better outcomes.
Change From Baseline in Functional Assessment of Chronic Illness Therapy-fatigue (FACIT-F) Score by Visit Over Time Through Week 48 | Baseline; Up to Week 48
  Change From baseline in FACIT-F Score at Week 48 will be reported. The FACIT-F is a questionnaire that assesses self-reported tiredness, weakness, and difficulty conducting usual activities due to fatigue. The subscale consists of 13-item instrument to measure fatigue. Each of the 13 items has a set of five response categories: Not at all (=0), A little bit (=1), Somewhat (=2), Quite a bit (=3) and Very much (=4). A total FACIT-Fatigue subscale score is calculated as the sum of the 13 item scores (reserved scores [4 - score]) and ranges from 0 to 52, with a higher score indicating less fatigue. Positive changes from baseline indicate improvement of fatigue. Items are reverse scored when appropriate to provide a scale in which higher scores represent better functioning or less fatigue.
Change From Baseline in Work Productivity and Activity Impairment Questionnaire: Crohn's Disease (WPAI:CD) by Visit Over Time Through Week 48 | Baseline; Up to Week 48
  Change from baseline in WPAI:CD by visit over time through Week 48 will be reported. The WPAI:CD assesses the impact of CD on work and activity during the past 7 days. The specificity of WPAI:CD is achieved by replacing "health problems" in the general health version of the WPAI with "CD." It consists of 6 questions, which elicit the following information: employment status; hours missed due to CD; hours missed due to other reasons; hours actually worked; the degree to which CD affected productivity while working from 0 (no effect) to 10 (maximum impairment); and the degree to which CD affected regular activities (from 0-10). The sum of worktime missed and impairment at work yields the overall work impairment (productivity loss) score; scores are expressed as percent of impairment/productivity loss, with higher scores indicating greater impairment.
Change from Baseline in Quality-of-life as Assessed by European Quality-of-Life Five Dimension Five Level Scale (EQ5D-5L) Score by Visit Over Time Through Week 48 | Baseline up to Week 48
  Change from baseline in quality-of-life (EQ5D-5L) score by visit over time through Week 48 will be reported. The EQ-5D-5L is a generic measure of health status. The EQ-5D-5L is a 5-item questionnaire that assesses 5 domains ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Change from Baseline in the Jorge-Wexner Score by Visit Over Time Through Week 48 | Baseline; Through Week 48
  Change from baseline in the Jorge-Wexner score by visit over time through Week 48 will be reported. The Jorge-Wexner scoring system cross-tabulates frequencies and different anal incontinence presentations.
Change from Baseline in the Inflammatory Bowel Disease-Disability Index (IBD-DI) by Visit Over Time Through Week 48 | Baseline; Through Week 48
  Change from baseline in the Inflammatory Bowel Disease-Disability Index (IBD-DI) by visit over time through Week 48 will be reported. The IBD-DI consists of 28 items that evaluate the 5 domains of overall health, body function, body structures, activity participation and environmental factors. Each item response is graded from 0 to 4 for each area evaluated (0 = very good; 1 = Good; 2 = medium; 3 = Bad; 4 = Very bad). The final composite score representative of the overall degree of disability ranging from -80 (maximum degree of disability) to 22 (no disability).
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to Week 48 and Week 96
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants with Treatment-emergent Serious Adverse Events (TESAEs) | Up to Week 48 and Week 96
  An serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product. TESAEs are defined as serious events between administration of study drug and after the last dose that were absent before treatment or that worsen relative to pretreatment state.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (151):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Gastroenterology Group Of Naples, Naples, Florida
  - AdventHealth Medical Group Blood & Marrow Transplant at Orlando, Orlando, Florida
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Washington University School Of Medicine, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - Digestive Disease Specialists Inc, Oklahoma City, Oklahoma
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Tyler Research Institute, LLC, Tyler, Texas
  - Swedish Medical Center, Seattle, Washington
- Australia (9):
  - Flinders Medical Centre, Adelaide
  - St Vincent's Hospital - Melbourne, Fitzroy
  - Liverpool Hospital, Liverpool
  - Fiona Stanley Hospital, Murdoch
  - Royal Prince Alfred Hospital, Newtown
  - Royal Adelaide Hospital, North Terrace
  - Royal Melbourne Hospital, Parkville
  - Royal Perth Hospital, Perth
  - Mater Hospital, South Brisbane
- Belgium (4):
  - Hopital Erasme, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Leuven, Leuven
  - CHU Sart Tilman, Liège
- Canada (5):
  - University of Alberta- Ziedler Ledcor Centre, Edmonton, Alberta
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Czechia (2):
  - Nemocnice Ceske Budejovice a s, České Budějovice
  - ISCARE a.s., Prague
- Egypt (4):
  - Alexandria University Hospital, Alexandria
  - National Hepatology and Tropical Medicine Research Institute, Cairo
  - Ain Shams University Hospital, Cairo
  - Cairo university, Giza
- France (6):
  - Clinique Ambroise Pare, Neuilly-sur-Seine
  - CHU de Nice Hopital de l Archet, Nice
  - Hopital Saint Joseph, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHRU Hopital de Pontchaillou, Rennes
  - CHRU Nancy Brabois, Vandœuvre-lès-Nancy
- Germany (5):
  - Charite - Campus Mitte, Berlin
  - JWG-University Hospital, Frankfurt
  - Universitatsklinikum Schleswig Holstein Kiel, Kiel
  - Universitaetsklinikum Mannheim, Mannheim
  - Universitaetsklinikum Ulm, Ulm
- Greece (8):
  - Evangelismos General Hospital of Athens, Athens
  - Hippokration Hospital, Athens
  - Sotiria General State Hospital of Chest Diseases, Athens
  - Alexandra General Hospital of Athens, Athens Attica
  - University Hospital of Heraklion, Heraklion
  - University Hospital Of Larissa, Larissa
  - Patras University Hospital, Pátrai
  - Hippokration Hospital, Thessaloniki
- Hungary (4):
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Semmelweis Egyetem, Budapest
  - Pecsi Tudomanyegyetem Orvostudomanyi Es Egeszsegtudomanyi Centrum, I. Belgyogyaszati Klinika, Pécs
  - Szegedi Tud Egyetem Szent Gyorgyi Albert Klin Kozp, Szeged
- Israel (4):
  - Haemek Medical Center, Afula
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center Beilinson Campus, Petah Tikva
- Italy (7):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale Classificato Equiparato Sacro Cuore Don Calabria di Negrar, Negrar ( Ve)
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Azienda Ospedaliera G.Salvini Ospedale di Rho, Rho
  - Policlinico Universitario Agostino Gemelli, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Japan (25):
  - KOKIKAI Tokatsu Tsujinaka Hospital, Abiko
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Hospital of the University of Occupational and Enviromental Health, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Kitakyushu Municipal Medical Center, Fukuoka-ken
  - Hiroshima University Hospital, Hiroshima
  - Sameshima Hospital, Kagoshima
  - Nara Medical University Hospital, Kashihara
  - Tsujinaka Hospital Kashiwanoha, Kashiwa
  - Nagasaki University Hospital, Nagasaki
  - Kojunkai Daido Clinic, Nagoya
  - Nagoya University Hospital, Nagoya
  - The Hospital of Hyogo College of Medicine, Nishinomiya
  - Okayama University Hospital, Okayama
  - Kinshukai Infusion Clinic, Osaka
  - JOHAS Osaka Rosai Hospital, Sakai
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - Tokyo Yamate Medical Center, Shinjuku-ku
  - Matsuda Hospital, Shizuoka
  - Osaka University Hospital, Suita
  - Kyorin University Hospital, Tokyo
  - Ieda Hospital, Toyota
  - Mie University Hospital, Tsu
  - Yokkaichi Hazu Medical Center, Yokkaichi
  - Yokohama Municipal Citizen's Hospital, Yokohama
- Jordan (5):
  - The Speciality Hospital (TSH) / Advanced Clinical Center, Amman
  - Jordan University Hospital, Amman
  - Abdali Hospital, Amman
  - Irbid Specialty Hospital, Irbid
  - King Abdullah University Hospital, Irbid
- Netherlands (4):
  - Academisch Medisch Centrum Universiteit van Amsterdam, Amsterdam
  - Radboudumc, Nijmegen
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht
- Poland (9):
  - Gastromed Kralisz Romatowski Stachurska Sp. j., Bialystok
  - Centrum Medyczne Promed, Krakow
  - Centrum Medyczne Med Gastr, Lodz
  - Centrum Medyczne Medyk, Rzeszów
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - GASTROMED Kopon Zmudzinski i wspolnicy SP j Specjalistyczne Centrum Gastrologii i Endoskopii, Torun
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Melita Medical Sp. z o.o., Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
- Portugal (3):
  - Uls Braga - Hosp. Braga, Braga
  - Uls Sao Jose - Hosp. Sto Antonio Dos Capuchos, Lisbon
  - H. Santo António - Centro Hospitalar do Porto, Porto
- Saudi Arabia (4):
  - King Fahad Specialist hospital, Dammam
  - King Abdulaziz Medical City, Jeddah
  - King Saud University Medical City, Riyadh
  - King Faisal Specialist Hospital & Research Center, Riyadh
- South Korea (5):
  - Inje University Haeundae Paik Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
- Spain (8):
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Arquitecto Marcide, Ferrol
  - Hosp. Univ. Dr. Josep Trueta, Girona
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Majadahonda
  - Hosp. Virgen Macarena, Seville
  - Hosp. Alvaro Cunqueiro, Vigo
  - Hosp. Univ. Miguel Servet, Zaragoza
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan
- Turkey (Türkiye) (5):
  - Gazi University Medical Faculty, Ankara
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Acibadem Kozyatagi Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
  - Mersin University Medical Faculty Hospital, Mersin
- United Kingdom (6):
  - Hull University Teaching Hospitals NHS Trust, Hull
  - London North West University Healthcare NHS Trust, London
  - Guys and St Thomas NHS Foundation Trust, London
  - St Georges University Hospital NHS Foundation Trust, London
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Pennine Acute Hospitals NHS Trust, Salford

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency